CLINICAL TRIAL: NCT06712927
Title: A Multicenter, Phase II Trial of Relatlimab, Nivolumab, and Ipilimumab in Patients With Asymptomatic and Symptomatic Melanoma Brain Metastases
Brief Title: Trial of Relatlimab, Nivolumab, and Ipilimumab in Patients With Asymptomatic and Symptomatic Melanoma Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-78364
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Melanoma; Brain Metastases
Keywords: Relatlimab; Nivolumab; Ipilimumab
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Ipilimumab; Nivolumab; Opdualag

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Asymptomatic (Experimental)
  Interventions: Drug: Ipilimumab; Drug: Nivolumab + Relatlimab FDC
- Cohort B: Symptomatic (Experimental)
  Interventions: Drug: Ipilimumab; Drug: Nivolumab + Relatlimab FDC

INTERVENTIONS:
Drug: Ipilimumab — 1 mg/kg of Ipilimumab will be administered via IV every 8 weeks. Participants will be assigned to Cohort A or B as per eligibility criteria. No randomization or blinding will occur
  Other Names: Yervoy
Drug: Nivolumab + Relatlimab FDC — Relatlimab 160mg + Nivo 480mg will be administered via IV every 4 weeks. Participants will be assigned to Cohort A or B as per eligibility criteria. No randomization or blinding will occur
  Other Names: Opdualag

SUMMARY:
This is a multicenter, phase II trial of relatlimab (rela), nivolumab (nivo), and ipilimumab (ipi) in patients with asymptomatic and symptomatic melanoma brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-uveal melanoma that has metastasized to the brain. At least 1 measurable intracranial target lesion (5-40mm) which was not previously treated with local therapy (no prior SRS to this lesion). Prior surgery for a brain metastasis is allowed but this lesion cannot be a target lesion.

   a. Growth or change in a lesion previously irradiated will not be considered measurable. Regrowth in cavity of previously excised lesion will not be considered measurable.
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 for Cohort A (asymptomatic), ECOG performance status 0-2 for Cohort B (symptomatic)
4. No prior anti-CTLA-4, anti-PD-1, or anti-LAG-3 therapy for unresectable stage III/IV melanoma. Prior CTLA-4, PD-1, and/or LAG-3 therapy in the neoadjuvant or adjuvant setting is acceptable if >6 months since last treatment. Participants may have had prior BRAF+MEK inhibitors for adjuvant therapy and/or unresectable/metastatic melanoma if >2 weeks have elapsed since last treatment.
5. Adequate organ function as assessed by the following parameters:

   1. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal (≤ 3 ×ULN); patients with liver metastasis ≤ 5 × ULN
   2. Estimated creatinine clearance (eCrCl) ≥ 30 mL/min using the Cockcroft-Gault formula at Screening
   3. Total bilirubin ≤ 1.5x ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels >1.5x ULN
6. Patients must have recovered from all prior anti-cancer therapy-related adverse events (AEs) to ≤ Grade 1 (per Common Terminology Criteria for Adverse Events [CTCAE] v 5.0), except for alopecia, vitiligo, thyroid dysfunction, hypophysitis, or adrenal insufficiency, prior to enrollment.
7. Cohort A (asymptomatic): participants must be free of neurologic signs and symptoms related to metastatic brain lesions and must not have required or received systemic corticosteroid therapy greater than physiologic replacement (>10 mg of prednisone/day or equivalent) in the 10 days prior to beginning protocol therapy. Cohort B (symptomatic): participants may be on steroids with doses no higher than a total daily dose of 4 mg of dexamethasone or equivalent that is stable or tapering within 10 days prior to treatment. Patients who are symptomatic and are not being treated with steroids are also eligible.
8. Participants with known human immunodeficiency virus (HIV)-infection are eligible providing they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 90 days prior to treatment.
9. Participants with a known history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection must have been treated and cured. Participants with HBV or HCV infection who are currently on treatment must have an undetectable HCV viral load prior to treatment.
10. Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (blocks are preferred) OR at least 4 unstained slides, with an associated pathology report, for testing of tumor PD-L1 expression:

    1. Tumor tissue should be of good quality based on total and viable tumor content.
    2. Patients who do not have tissue specimens may undergo a biopsy during the screening period. Acceptable samples include core-needle biopsies for deep tumor tissue or excisional, incisional, punch, or forceps biopsies for cutaneous, subcutaneous, or mucosal lesions. Fine Needle Aspirations (FNA) will not be considered acceptable for tissue procurement.
    3. Tumor tissue from bone metastases is not evaluable for PD-L1 expression and is therefore not acceptable.
    4. However, if repeat biopsy is not feasible, and no archival tissue available patient still may be enrolled.
11. Any radiation treatment or excision of non-target brain lesions must have occurred ≥ 1 weeks before the start of dosing for this study. NOTE: The radiation field must not have included the brain index lesion(s).
12. Radiation to non-CNS lesions is allowed and does not require a washout period for treatment initiation. Any radiation-related toxicity must have recovered to ≤ Grade 1 (per Common Terminology Criteria for Adverse Events [CTCAE] v 5.0).
13. Women of child-bearing potential (WOCBP) must not be breastfeeding and must have a negative pregnancy test within 3 days prior to initiation of dosing. WOCBP (or female partners of male participants) must agree to use an acceptable method of birth control from the time of the negative pregnancy test, through the duration of treatment with the study combination and for 12 months after their last dose of any study component medication.

    NOTE: A female participant is eligible to participate if she is not a woman of childbearing potential.

    Approved methods of birth control are as follows:

    Combined (estrogen and progesterone containing) hormonal birth control associated with inhibition of ovulation: oral, intravaginal, transdermal Progesterone-only hormonal birth control associated with inhibition of ovulation: oral, injectable, implantable Intrauterine device (IUD) Intrauterine hormone-releasing system (IUS) Bilateral tubal occlusion Vasectomized partner True sexual abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar ovulation, symptothermal, post-ovulation methods) is not acceptable
14. Patients (or legally authorized representative) must have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an ICF approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC) and agree to abide by the study restrictions and return to the site for the required assessments.

Exclusion Criteria

1. Another primary malignancy within the previous 3 years (with the exception of carcinoma in situ of the breast, cervix, or bladder; localized prostate cancer; and non-melanoma skin cancer that has been adequately treated).
2. Active medical illness(es) that would pose increased risk for study participation, including: active systemic infections (including COVID-19), coagulation disorders, or other major active medical illnesses of the cardiovascular, respiratory, or immune systems.
3. Active autoimmune disease that has required systemic therapy with corticosteroids or other immunosuppressive agents within the past 3 years (excluding immune-related adverse events from immunotherapy as described above.
4. Implanted device that precludes the use of MRI.
5. Prior Grade 4 treatment-related AE with immune checkpoint inhibitor treatment.
6. History of leptomeningeal metastasis determined by imaging or lumbar puncture.
7. Prior whole brain radiation therapy (WBRT)
8. Women who are breast-feeding or pregnant
9. History of clinically significant cardiac disease or congestive heart failure > New York Heart Association (NYHA) class 2. Subjects must not have unstable angina (anginal symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months or a history of myocarditis
10. Troponin T (TnT) or I (TnI) > 2 × institutional ULN. Participants with TnT or TnI levels between > 1 to 2 × ULN will be permitted if repeat levels within 24 hours are ≤ 1 ULN. If TnT or TnI levels are between >1 to 2 × ULN within 24 hours, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 × ULN, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. Notification of the decision to enroll the participant following cardiologist recommendation has to be made to the principal investigator.
11. Investigational drug use within 14 days (or 5 half-lives, whichever is longer) of the first dose of study treatment.
12. Dexamethasone use > 4mg/day (or equivalent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Intracranial clinical benefit rate | 6 months
  Intracranial clinical benefit rate, defined as the percentage of patients who had a complete response (CR), partial response (PR), or stable disease for at least 6 months per modified RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Evaluation of Safety and Adverse Events Using CTCAE v5.0 | 6 months
  Safety will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Extracranial objective response rate | 6 months
  Extracranial objective response rate, defined as the percentage of patients who had a complete response (CR) or partial response (PR) per RECIST 1.1 criteria.
Global objective response rate | 6 months
  Global objective response rate, defined as the percentage of patients who had a complete response (CR) or partial response (PR) per modified RECIST 1.1 criteria.
Extracranial clinical benefit rate | 6 months
  Extracranial clinical benefit rate, defined as the percentage of patients who had a complete response (CR), partial response (PR), or stable disease for at least 6 months per RECIST 1.1 criteria.
Global clinical benefit rate | 6 months
  Global clinical benefit rate, defined as the percentage of patients who had a complete response (CR), partial response (PR), or stable disease for at least 6 months per modified RECIST 1.1 criteria.
Duration of response | 60 months
  Duration of response, measured from time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started) or death.
Progression-free survival | 60 months
  Progression-free survival, defined as the duration of time from start of treatment to time of progression or death.
Intracranial progression-free survival | 60 month
  Intracranial progression-free survival, defined as the duration of time from start of treatment to time of intracranial progression or death.
Overall survival | 60 months
  Overall survival, defined as the duration of time from the start of treatment to death.
Intracranial Objective response rate | 6 months
  Intracranial objective response rate, defined as the percentage of patients who had a complete response (CR) or partial response (PR) per modified RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Allison B Warner, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States